CLINICAL TRIAL: NCT05039424
Title: A Randomized, Sham-controlled Trial: Endoscopic Myotomy of the Pylorus To Improve Emptying and Symptoms (EMPTIES)
Brief Title: Endoscopic Myotomy of the Pylorus To Improve Emptying and Symptoms Trial
Acronym: EMPTIES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Allemang (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Matthew Allemang, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-160; 5R01DK120830-02 (NIH)
Record Dates: First submitted 2021-08-19; First posted 2021-09-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy; Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: A comparative effectiveness, single center (with two surgical units), randomized (1:1) study of POP vs. sham endoscopic surveillance in patients with medically refractory gastroparesis. This study will also include a crossover approach, offering POP to patients randomized to the sham arm, if they remain symptomatic at 12 weeks post randomization.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic per-oral pyloromyotomy (POP) (Active Comparator): Participants will undergo Endoscopic per-oral pyloromyotomy (POP).
  Interventions: Procedure: Endoscopic per-oral pyloromyotomy (POP)
- Sham / Control Arm (Sham Comparator): Participants will undergo a diagnostic esophagogastroduodenoscopy (EGD) without pyloric disruption. Following the 12-week blinded trial period, these participants will be unblinded and offered Endoscopic per-oral pyloromyotomy (POP) if they remain symptomatic.
  Interventions: Procedure: Endoscopic per-oral pyloromyotomy (POP); Procedure: Diagnostic esophagogastroduodenoscopy (EGD) without pyloric disruption

INTERVENTIONS:
Procedure: Endoscopic per-oral pyloromyotomy (POP) — Per-oral pyloromyotomy (POP), alternatively knows as gastric per-oral endoscopic myotomy (G-POEM), accomplishes longitudinal division of the pylorus using an endoscope. This procedure involves utilizing endoscopic electrosurgical knife to make an incision in the gastric mucosa and develop a submucosal tunnel to visualize the pyloric ring. The pyloric ring is divided longitudinally, and the mucosotomy incision is sealed with endoscopic clips.
Procedure: Diagnostic esophagogastroduodenoscopy (EGD) without pyloric disruption — While under general anesthesia, a standard gastroscope is introduced and a diagnostic upper endoscopy is performed. The operator talks through the procedure steps as if completing POP. The gastroscope is withdrawn and the patient is extubated.
  Arms: Sham / Control Arm

SUMMARY:
A randomized clinical trial comparing endoscopic per-oral pyloromyotomy (POP) versus a control sham intervention (diagnostic esophagogastroduodenoscopy (EGD) without pyloric disruption) in patients with medically refractory gastroparesis.

DETAILED DESCRIPTION:
A comparative effectiveness, single center (with two surgical units), randomized (1:1) study of endoscopic per-oral pyloromyotomy (POP) versus a control sham intervention (diagnostic esophagogastroduodenoscopy (EGD) without pyloric disruption) in adult patients with medically refractory gastroparesis who have failed management with dietary, lifestyle, and pharmacological therapy for at least six months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75
2. Diagnosis of medically refractory gastroparesis by 4 hour non-extrapolated solid phase gastric emptying study completed within 12 months of enrollment. Medical refractoriness is defined by at least 6 months of medical treatment with no significant improvement in baseline symptoms
3. Completion of all routine assessments in our multidisciplinary gastroparesis clinic, which includes evaluation by gastroenterology, behavioral health, and nutrition specialists
4. Ability to take oral medication and be willing to adhere to the post-procedure dietary and medication regimen
5. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation
6. Stated willingness to comply with all study procedures and availability for the duration of the study
7. Willingness and reasonable expectation that the individual will be able to travel to the study site for the intervention and each scheduled in-person assessment, as well as virtual assessments if necessary
8. Be able to speak and read the English language.

Exclusion Criteria:

1. Active use of narcotic pain medication
2. Presence of concomitant gastrointestinal transit disorder such as small bowel dysmotility or uncontrolled colonic dysmotility (As defined by clinical judgement or < 3 bowel movements per week)
3. Etiology of gastroparesis is post-surgical
4. Pregnancy or lactation
5. History of egg allergy
6. Prior surgical intervention of the stomach or gastric pylorus
7. Current parenteral nutrition
8. Uncontrolled coagulopathy (platelet count <50,000 and INR>1.5) or use of anticoagulant medications (with the exception of antiplatelet therapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index (GCSI) | Baseline, 12 weeks post-procedure
  Change in Gastroparesis Cardinal Symptom Index (GCSI) at Baseline to 12 weeks post-procedure. Possible scores range from 0 (None) to 5 (Very Severe).

SECONDARY OUTCOMES:
Gastric Emptying | Baseline, 12 weeks post-procedure
  Change in gastric emptying as measured by a standardized 4-hour solid scintigraphic gastric emptying study at Baseline to 12 weeks post-procedure
36-Item Short Form; Quality of Life Survey | Baseline,12 weeks post-procedure
  Change in 36-Item Short Form Survey (SF-36) score from Baseline to 12 weeks post-procedure. The weighted sums of responses to questions in the survey produce eight separate scales which are scored from 0-100, with zero indication maximum disability and one hundred indicating no disability in that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Allemang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasler WL. Gastroparesis: symptoms, evaluation, and treatment. Gastroenterol Clin North Am. 2007 Sep;36(3):619-47, ix. doi: 10.1016/j.gtc.2007.07.004. PMID 17950441
- [Background] Wang YR, Fisher RS, Parkman HP. Gastroparesis-related hospitalizations in the United States: trends, characteristics, and outcomes, 1995-2004. Am J Gastroenterol. 2008 Feb;103(2):313-22. doi: 10.1111/j.1572-0241.2007.01658.x. Epub 2007 Nov 28. PMID 18047541
- [Background] Mayer-Davis EJ, Lawrence JM, Dabelea D, Divers J, Isom S, Dolan L, Imperatore G, Linder B, Marcovina S, Pettitt DJ, Pihoker C, Saydah S, Wagenknecht L; SEARCH for Diabetes in Youth Study. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Apr 13;376(15):1419-1429. doi: 10.1056/NEJMoa1610187. PMID 28402773
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Gastroparesis Cardinal Symptom Index (GCSI): development and validation of a patient reported assessment of severity of gastroparesis symptoms. Qual Life Res. 2004 May;13(4):833-44. doi: 10.1023/B:QURE.0000021689.86296.e4. PMID 15129893
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Background] Abell TL, Bernstein RK, Cutts T, Farrugia G, Forster J, Hasler WL, McCallum RW, Olden KW, Parkman HP, Parrish CR, Pasricha PJ, Prather CM, Soffer EE, Twillman R, Vinik AI. Treatment of gastroparesis: a multidisciplinary clinical review. Neurogastroenterol Motil. 2006 Apr;18(4):263-83. doi: 10.1111/j.1365-2982.2006.00760.x. PMID 16553582
- [Background] Yu D, Ramsey FV, Norton WF, Norton N, Schneck S, Gaetano T, Parkman HP. The Burdens, Concerns, and Quality of Life of Patients with Gastroparesis. Dig Dis Sci. 2017 Apr;62(4):879-893. doi: 10.1007/s10620-017-4456-7. Epub 2017 Jan 21. PMID 28110376
- [Background] Lacy BE, Crowell MD, Mathis C, Bauer D, Heinberg LJ. Gastroparesis: Quality of Life and Health Care Utilization. J Clin Gastroenterol. 2018 Jan;52(1):20-24. doi: 10.1097/MCG.0000000000000728. PMID 27775961
- [Background] Jones MP, Maganti K. A systematic review of surgical therapy for gastroparesis. Am J Gastroenterol. 2003 Oct;98(10):2122-9. doi: 10.1111/j.1572-0241.2003.07721.x. PMID 14572555
- [Background] Lal N, Livemore S, Dunne D, Khan I. Gastric Electrical Stimulation with the Enterra System: A Systematic Review. Gastroenterol Res Pract. 2015;2015:762972. doi: 10.1155/2015/762972. Epub 2015 Jul 12. PMID 26246804
- [Background] Ramkumar D, Schulze KS. The pylorus. Neurogastroenterol Motil. 2005 Jun;17 Suppl 1:22-30. doi: 10.1111/j.1365-2982.2005.00664.x. PMID 15836452
- [Background] Mearin F, Camilleri M, Malagelada JR. Pyloric dysfunction in diabetics with recurrent nausea and vomiting. Gastroenterology. 1986 Jun;90(6):1919-25. doi: 10.1016/0016-5085(86)90262-3. PMID 3699409
- [Background] Koch KL, Calles-Escandon J. Diabetic gastroparesis. Gastroenterol Clin North Am. 2015 Mar;44(1):39-57. doi: 10.1016/j.gtc.2014.11.005. PMID 25667022
- [Background] Toro JP, Lytle NW, Patel AD, Davis SS Jr, Christie JA, Waring JP, Sweeney JF, Lin E. Efficacy of laparoscopic pyloroplasty for the treatment of gastroparesis. J Am Coll Surg. 2014 Apr;218(4):652-60. doi: 10.1016/j.jamcollsurg.2013.12.024. Epub 2013 Dec 24. PMID 24529808
- [Background] Hibbard ML, Dunst CM, Swanstrom LL. Laparoscopic and endoscopic pyloroplasty for gastroparesis results in sustained symptom improvement. J Gastrointest Surg. 2011 Sep;15(9):1513-9. doi: 10.1007/s11605-011-1607-6. Epub 2011 Jul 1. PMID 21720926
- [Background] Lebares C, Swanstrom LL. Per-Oral Pyloromyotomy (POP): An Emerging Application of Submucosal Tunneling for the Treatment of Refractory Gastroparesis. Gastrointest Endosc Clin N Am. 2016 Apr;26(2):257-270. doi: 10.1016/j.giec.2015.12.012. PMID 27036896
- [Background] Allemang MT, Strong AT, Haskins IN, Rodriguez J, Ponsky JL, Kroh M. How I Do It: Per-Oral Pyloromyotomy (POP). J Gastrointest Surg. 2017 Nov;21(11):1963-1968. doi: 10.1007/s11605-017-3510-2. Epub 2017 Jul 27. PMID 28752406
- [Background] Rodriguez JH, Haskins IN, Strong AT, Plescia RL, Allemang MT, Butler RS, Cline MS, El-Hayek K, Ponsky JL, Kroh MD. Per oral endoscopic pyloromyotomy for refractory gastroparesis: initial results from a single institution. Surg Endosc. 2017 Dec;31(12):5381-5388. doi: 10.1007/s00464-017-5619-5. Epub 2017 May 31. PMID 28567693
- [Background] Rodriguez J, Strong AT, Haskins IN, Landreneau JP, Allemang MT, El-Hayek K, Villamere J, Tu C, Cline MS, Kroh M, Ponsky JL. Per-oral Pyloromyotomy (POP) for Medically Refractory Gastroparesis: Short Term Results From the First 100 Patients at a High Volume Center. Ann Surg. 2018 Sep;268(3):421-430. doi: 10.1097/SLA.0000000000002927. PMID 30004920
- [Background] Woodhouse S, Hebbard G, Knowles SR. Psychological controversies in gastroparesis: A systematic review. World J Gastroenterol. 2017 Feb 21;23(7):1298-1309. doi: 10.3748/wjg.v23.i7.1298. PMID 28275310
- [Background] Soykan I, Sivri B, Sarosiek I, Kiernan B, McCallum RW. Demography, clinical characteristics, psychological and abuse profiles, treatment, and long-term follow-up of patients with gastroparesis. Dig Dis Sci. 1998 Nov;43(11):2398-404. doi: 10.1023/a:1026665728213. PMID 9824125
- [Background] Arts J, Holvoet L, Caenepeel P, Bisschops R, Sifrim D, Verbeke K, Janssens J, Tack J. Clinical trial: a randomized-controlled crossover study of intrapyloric injection of botulinum toxin in gastroparesis. Aliment Pharmacol Ther. 2007 Nov 1;26(9):1251-8. doi: 10.1111/j.1365-2036.2007.03467.x. PMID 17944739
- [Background] McCallum RW, Snape W, Brody F, Wo J, Parkman HP, Nowak T. Gastric electrical stimulation with Enterra therapy improves symptoms from diabetic gastroparesis in a prospective study. Clin Gastroenterol Hepatol. 2010 Nov;8(11):947-54; quiz e116. doi: 10.1016/j.cgh.2010.05.020. Epub 2010 Jun 9. PMID 20538073
- [Background] McCallum RW, Sarosiek I, Parkman HP, Snape W, Brody F, Wo J, Nowak T. Gastric electrical stimulation with Enterra therapy improves symptoms of idiopathic gastroparesis. Neurogastroenterol Motil. 2013 Oct;25(10):815-e636. doi: 10.1111/nmo.12185. Epub 2013 Jul 29. PMID 23895180
- [Background] Gonzalez JM, Benezech A, Vitton V, Barthet M. G-POEM with antro-pyloromyotomy for the treatment of refractory gastroparesis: mid-term follow-up and factors predicting outcome. Aliment Pharmacol Ther. 2017 Aug;46(3):364-370. doi: 10.1111/apt.14132. Epub 2017 May 15. PMID 28504312
- [Background] Mancini SA, Angelo JL, Peckler Z, Philp FH, Farah KF. Pyloroplasty for Refractory Gastroparesis. Am Surg. 2015 Jul;81(7):738-46. PMID 26140897
- [Background] Khashab MA, Ngamruengphong S, Carr-Locke D, Bapaye A, Benias PC, Serouya S, Dorwat S, Chaves DM, Artifon E, de Moura EG, Kumbhari V, Chavez YH, Bukhari M, Hajiyeva G, Ismail A, Chen YI, Chung H. Gastric per-oral endoscopic myotomy for refractory gastroparesis: results from the first multicenter study on endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2017 Jan;85(1):123-128. doi: 10.1016/j.gie.2016.06.048. Epub 2016 Jun 25. PMID 27354102
- [Background] Gersin KS, Rothstein RI, Rosenthal RJ, Stefanidis D, Deal SE, Kuwada TS, Laycock W, Adrales G, Vassiliou M, Szomstein S, Heller S, Joyce AM, Heiss F, Nepomnayshy D. Open-label, sham-controlled trial of an endoscopic duodenojejunal bypass liner for preoperative weight loss in bariatric surgery candidates. Gastrointest Endosc. 2010 May;71(6):976-82. doi: 10.1016/j.gie.2009.11.051. Epub 2010 Mar 20. PMID 20304396